CLINICAL TRIAL: NCT00105300
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study of the Human Anti-TNF Monoclonal Antibody Adalimumab for the Induction of Clinical Remission in Subjects With Moderate to Severe Crohn's Disease Who Have Lost Response or Are Intolerant to Infliximab
Brief Title: Study of the Human Anti-TNF Monoclonal Antibody Adalimumab for the Induction of Clinical Remission in Subjects With Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M04-691
Record Dates: First submitted 2005-03-11; First posted 2005-03-14 (Estimated); Last update posted 2006-08-15 (Estimated); Status verified 2006-08

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

INTERVENTIONS:
Drug: Adalimumab

SUMMARY:
The goal of this study is to test whether adalimumab can induce clinical remission in subjects with active Crohn's disease who have been initially treated with infliximab and either lost response or discontinued its use as a result of intolerance to the drug.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18 and 75 who are diagnosed with mild to moderate Crohn's disease (defined by a CDAI [Crohn's Disease Activity Index] score of 220 and 450)
* Normal lab parameters
* Are willing to give informed consent
* Have previously used and either were intolerant to or lost response to infliximab

Exclusion Criteria:

* History of certain types of cancer
* Diagnosis of ulcerative colitis
* Pregnant female or breast feeding subjects
* Known obstructive strictures
* Surgical bowel resection in the past 6 months
* History of listeria, human immunodeficiency virus (HIV), central nervous system demyelinating disease or untreated TB (tuberculosis)
* History of poorly controlled medical conditions
* Specific doses and durations of Crohn's medications
* Subjects that have previously used infliximab and have never clinically responded unless primary non-response was due to a treatment limiting reaction to infliximab

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-10

PRIMARY OUTCOMES:
Induction of clinical remission (CDAI score < 150 at Week 4)

SECONDARY OUTCOMES:
Clinical response measured as
Decrease in Baseline CDAI score >= 70 points at Week 4
Decrease in Baseline CDAI score >= 100 points at Week 4
Changes in IBDQ scores at Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information 1-800-633-9110, Study Director — Abbott
Locations (56):
- United States (46):
  - Clinical Research Associates, Huntsville, Alabama
  - Capitol Gastroenterology Consultants Medical Group, Inc., Roseville, California
  - Medical Associates Research Group, San Diego, California
  - Sharp Rees-Stealy Medical Group, San Diego, California
  - SMC-Trauma Research, Englewood, Colorado
  - Clinical Research of West Florida, Inc, Clearwater, Florida
  - V.A. Medical Center, Gainesville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Pinnacle Trials, Inc., Atlanta, Georgia
  - Atlanta Gastroenterology Assoc., Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - Ntouch Research, Peoria, Illinois
  - Outpatient Clinical Research Facility University of Indianapolis, Indianapolis, Indiana
  - University of Kentucky Medical Center Division of Digestive Diseases, Lexington, Kentucky
  - Drug Research Services, Inc., Metairie, Louisiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Charm City Research, Towson, Maryland
  - Minnesota Gastroenterology P.A., Plymouth, Minnesota
  - Mayo Clinic Research, Rochester, Minnesota
  - Gastrointestinal Associated, P.A., Jackson, Mississippi
  - Glen Gordon, MD, Mexico, Missouri
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Atlantic Gastroenterology Associates, LLC, Egg Harbor, New Jersey
  - Long Island Clinical Research Assoc. LLP, Great Neck, New York
  - NY Center for Clinical Research, Lake Success, New York
  - Mount Sinai School of Medicine IBD Research Center, New York, New York
  - Asheville Gastroenterology Associates, Ashville, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Gastrointestinal and Liver Disease Consultants, Dayton, Ohio
  - Gastroenterology Associates of Cleveland, Mayfield Heights, Ohio
  - The Oregon Clinic, PC Gastroenterology Division, Portland, Oregon
  - Regional Gastroenterologist Associates of Lancaster, Lancaster, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Columbia Gastro Associates, Columbia, South Carolina
  - Gastrointestinal Associates, Knoxville, Tennessee
  - Gastroenterology Center of the Mid South, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Austin Gastroenterology, Austin, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Internal Medicine Associates, Danville, Virginia
  - Digestive and Liver Disease, Norfolk, Virginia
  - Spokane Digestive Disease Center, Spokane, Washington
  - Discovery Research International, LLC, Milwaukee, Wisconsin
- Belgium (2):
  - Imelda Ziekenhuis, Bonheiden
  - UZ Gasthuisberg, Leuven
- Canada (7):
  - Heritage Medical Research Clinic Health Sciences Centre University of Calgary, Calgary, Alberta
  - Liver and Intestinal Disease Research Center, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Winnipeg Health Sciences Centre, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Toronto Digestive Disease Assoc. Inc, Toronto, Ontario
  - Royal Victoria Hospital, Montreal, Quebec
- Hopital Claude Claude Huriez Hospital, Lille, Cedex, France

REFERENCES:
- [Derived] Sandborn WJ, Rutgeerts P, Enns R, Hanauer SB, Colombel JF, Panaccione R, D'Haens G, Li J, Rosenfeld MR, Kent JD, Pollack PF. Adalimumab induction therapy for Crohn disease previously treated with infliximab: a randomized trial. Ann Intern Med. 2007 Jun 19;146(12):829-38. doi: 10.7326/0003-4819-146-12-200706190-00159. Epub 2007 Apr 30. PMID 17470824